CLINICAL TRIAL: NCT00099008
Title: Phase I Multiple Dose Clinical Study of Soy Isoflavones in Healthy, Post-Menopausal Women
Brief Title: Genistein in Preventing Breast or Endometrial Cancer in Healthy Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UNC-GCRC-2107; CDR0000393450 (Other: PDQ number)
Record Dates: First submitted 2004-12-08; First posted 2004-12-09 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Breast Cancer; Endometrial Cancer
Keywords: breast cancer; endometrial cancer
MeSH Terms: conditions — Breast Neoplasms; Endometrial Neoplasms | interventions — Genistein

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Genistein
  Interventions: Dietary Supplement: Genistein
- Arm II (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Genistein — oral Genistein twice daily on days 1-84
  Other Names: PTI G-2535
  Arms: Arm I
Dietary Supplement: Placebo — oral Placebo twice daily on days 1-84
  Arms: Arm II

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. The use of genistein may be effective in preventing breast or endometrial cancer.

PURPOSE: This randomized phase I trial is studying the effectiveness of genistein in preventing breast or endometrial cancer in healthy postmenopausal women.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effects of genistein vs placebo on DNA damage and apoptosis by conducting COMET, TUNEL, Caspase-3, and AP site assays in healthy postmenopausal women.
* Compare the effects of these drugs on gene expression in an estrogen-sensitive tissue by oligoarray profiling in these participants.
* Determine the effect of genistein on estrogenic effects by self-reported side effects, measurement of sex hormone-binding globulin, follicle-stimulating hormone, luteinizing hormone, and estrogen levels, and expression of known estrogen-sensitive genes in these participants.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Participants are stratified according to their study ID numbers. Participants are randomized to 1 of 2 treatment arms.

* Arm I: Participants receive oral genistein twice daily on days 1-84.
* Arm II: Participants receive oral placebo twice daily on days 1-84. In both arms, treatment continues in the absence of dysplasia, malignancy, unacceptable toxicity, or gross noncompliance.

Participants are followed at days 7, 14, 28, 56, and 84 during study treatment and at day 28 after completion of study treatment.

PROJECTED ACCRUAL: A total of 30 participants (20 for arm I and 10 for arm II) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Healthy participants

  * Papanicolaou test (pap smear) normal within the past 13 months
  * Mammogram normal within the past 13 months
* No history of breast cancer
* Not at high-risk (5-year risk < 1.9%) for breast cancer according to NCI's Breast Cancer Risk Assessment Tool
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 45 to 70

Sex

* Female

Menopausal status

* Postmenopausal

  * Last spontaneous menstrual bleeding > 12 months ago

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC ≥ 3,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 2.0 mg/dL
* ALT and AST < 2 times normal
* No significant abnormality of the liver by physical exam

Renal

* Creatinine < 2.0 mg/dL

Cardiovascular

* No significant cardiac disease
* No New York Heart Association class III or IV heart disease
* No significant abnormality of the heart by physical exam

Pulmonary

* No significant abnormality of the lung by physical exam

Other

* Body mass index < 35
* Follicle-stimulating hormone > 27 mIU/mL
* Thyroid or endocrine function test normal
* Alcohol intake ≤ 2 drinks/day or ≤14 drinks/week
* Not pregnant
* No intermediate equol values (≥10 ug/L to ≤ 20 ug/L) on soy challenge
* No history of seizures
* No significant abnormality of the spleen or other abdominal organs by physical exam
* No neurologic abnormality by physical exam
* No significant metabolic abnormality on the biochemical screen
* No history of substance abuse or addiction
* No tobacco use
* No diets containing > 20 mg of genistein/day or > 40 mg isoflavone/day
* No known intolerance to soy
* No other serious medical illness
* No active malignancy or malignancy initially diagnosed within the past 2 years except curatively treated nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 2 years since prior chemotherapy
* No concurrent chemotherapy

Endocrine therapy

* More than 3 months since prior hormonal or estrogen therapy
* More than 3 months since prior tamoxifen or other selective estrogen-receptor modulators
* More than 1 month since prior supplements containing phytoestrogens or that have estrogenic side effects (soy isoflavones or PC-SPECS)
* No concurrent thyroid medication

  * Other concurrent endocrine medication allowed provided medication was initiated ≥ 3 months before study entry AND participant has been on a stable regimen for the past 3 months

Radiotherapy

* Not specified

Surgery

* No prior hysterectomy or oophorectomy

Other

* More than 3 months since prior antibiotics

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-03; Primary Completion 2005-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Efficacy of genistein on DNA and apoptosis | 112 days
  Compare the effects of genistein vs placebo on DNA damage and apoptosis by conducting COMET, TUNEL, Caspase-3, and AP site assays in healthy postmenopausal women.

CONTACTS AND LOCATIONS:
Overall Officials: Steven H. Zeisel, MD, PhD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Result] Pop EA, Fischer LM, Coan AD, Gitzinger M, Nakamura J, Zeisel SH. Effects of a high daily dose of soy isoflavones on DNA damage, apoptosis, and estrogenic outcomes in healthy postmenopausal women: a phase I clinical trial. Menopause. 2008 Jul-Aug;15(4 Pt 1):684-92. doi: 10.1097/gme.0b013e318167b8f2. PMID 18446090